CLINICAL TRIAL: NCT00320593
Title: Correction of Myopia Evaluation Trial 2 (COMET2): A Randomized Trial of the Effect of Progressive Addition Lenses Versus Single Vision Lenses on Low Myopia Associated With Large Accommodative Lags and Near Esophoria in Children
Brief Title: Correction of Myopia Evaluation Trial 2
Acronym: COMET2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEI-123; 2U10EY011751 (NIH); 5U10EY011751 (NIH)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Myopia
Keywords: Myopia; Progressive Addition Lenses (PALs); Single Vision Lenses (SVLs); Accommodative lags; Near esophoria; Refractive error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progressive addition lenses (PALs) (Active Comparator): Varilux Ellipse progressive addition lenses (PALs) with a +2.00 D addition
  Interventions: Device: Progressive Addition Lenses (PALs)
- Single vision lenses (SVLs) (Active Comparator): Single vision lenses
  Interventions: Device: Single Vision Lenses (SVLs)

INTERVENTIONS:
Device: Progressive Addition Lenses (PALs) — Varilux Ellipse progressive addition lenses (PALs) with a +2.00 D addition
  Arms: Progressive addition lenses (PALs)
Device: Single Vision Lenses (SVLs) — Single vision lenses
  Arms: Single vision lenses (SVLs)

SUMMARY:
The purpose of the study is to determine if progressive addition lenses (PALs) versus single vision lenses (SVLs) slow the progression of low myopia in children with poor accommodative responses (i.e., large accommodative lags) and near esophoria.

DETAILED DESCRIPTION:
Myopia is a significant public health problem that affects at least 34% of children in the United States and a much higher percentage in Asia. It is a predisposing factor for retinal detachment, myopic retinopathy, and glaucoma, thus contributing to loss of vision and blindness. As might be expected for such a prevalent condition, treatment costs are high. If interventions to retard myopia progression are successful, sight-threatening complications might be avoided and costs should be reduced.

The study has been designed as a simple trial that, other than the type of lenses being determined through the randomization process and the addition of accommodation testing using an autorefractor, largely approximates standard clinical practice.

Screening consists of non-cycloplegic procedures of subjective refraction, testing of oculomotor alignment, and testing of accommodative response using the Grand Seiko autorefractor.

Patients who appear to be eligible for the randomized trial will be tested with their eyes dilated to determine whether refractive error in each eye is within the eligibility range for the randomized trial. Patients will be randomized to either progressive addition lenses (PALs) with a +2.00 D addition or to single vision lenses (SVLs). Children will have three years of follow up, with visits every 6 months.

The primary outcome visit is timed 3 years from randomization, with the primary analysis being a comparison of the average change from baseline to 3 years in amount of myopia between children in the single-vision lens group and the children in the progressive-addition lens group. The primary outcome is change in spherical equivalent refractive error (SER) in diopters (D) as measured by cycloplegic autorefraction.

A separate ancillary study nested within the screening process will collect data on two additional methods of measuring accommodation, Monocular Estimate Method (MEM) retinoscopy and Nott retinoscopy. The aim of the ancillary study to help determine whether a simple, effective measure exists that can be easily used by clinicians to identify children with reduced accommodative response who, if they have low myopia and esophoria, might benefit from the treatment with PALs.

ELIGIBILITY:
Inclusion Criteria:

* Refractive error determined by cycloplegic autorefraction which meets all of the following:

  1. Spherical equivalent: -0.50 to -3.00 D in both eyes
  2. Astigmatism <= 1.5 D in both eyes
  3. Anisometropia <= 1.00 D difference between eyes in spherical equivalent
* Visual acuity is at least 20/20 with best subjective refraction in both eyes
* Accommodative response at near (33 cm) is less than 2.0D by non-cycloplegic autorefraction
* Near esophoria (>= 2.0 PD) present by alternate prism and cover test (APCT) at near using best refractive correction determined from non-cycloplegic subjective refraction

Exclusion Criteria:

* Strabismus present by cover-uncover test at far, near, and/or near with +2.00D over best subjective refraction
* Current or prior use of PALs, bifocals, or contact lenses in either eye (prior or current use of SVLs is allowed)

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2005-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Gwiazda, Ph.D., Study Chair — New England College of Optometry; Wendy L Marsh-Tootle, Principal Investigator — University of Alabama at Birmingham School of Optometry; Ruth E Manny, Principal Investigator — University of Houston College of Optometry; Erik M Weissberg, Principal Investigator — New England College of Optometry; David I Silbert, Principal Investigator — Family Eye Group; Don W Lyon, Principal Investigator — Indiana University; Mitchell M Scheiman, Principal Investigator — Pennsylvania College of Optometry; Marjean T Kulp, Principal Investigator — Ohio State University; Susan A Cotter, Principal Investigator — Southern California College of Optometry at Marshall B. Ketchum University
Locations (8):
- United States (8):
  - University of Alabama- Birmingham, School of Optometry, Birmingham, Alabama
  - Southern California College of Optometry, Fullerton, California
  - Indiana School of Optometry, Bloomington, Indiana
  - New England College of Optometry, Boston, Massachusetts
  - Ohio State University College of Optometry, Columbus, Ohio
  - Family Eye Group, Lancaster, Pennsylvania
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - University of Houston College of Optometry, Houston, Texas

REFERENCES:
- [Result] Correction of Myopia Evaluation Trial 2 Study Group for the Pediatric Eye Disease Investigator Group; Manny RE, Chandler DL, Scheiman MM, Gwiazda JE, Cotter SA, Everett DF, Holmes JM, Hyman LG, Kulp MT, Lyon DW, Marsh-Tootle W, Matta N, Melia BM, Norton TT, Repka MX, Silbert DI, Weissberg EM. Accommodative lag by autorefraction and two dynamic retinoscopy methods. Optom Vis Sci. 2009 Mar;86(3):233-43. doi: 10.1097/OPX.0b013e318197180c. PMID 19214130
- [Result] Correction of Myopia Evaluation Trial 2 Study Group for the Pediatric Eye Disease Investigator Group. Progressive-addition lenses versus single-vision lenses for slowing progression of myopia in children with high accommodative lag and near esophoria. Invest Ophthalmol Vis Sci. 2011 Apr 25;52(5):2749-57. doi: 10.1167/iovs.10-6631. PMID 21282579
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2005 and March 2007, 118 subjects age 8 to <12 years were enrolled in the study at 8 clinical centers.
Groups:
- Single Vision Lenses (SVLs): Standard single vision lenses
Period: Overall Study
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Started | 59 | 59
Completed | 52 (Completed defined as completing the 3 year primary outcome exam) | 58 (Completed defined as completing the 3 year primary outcome exam)
Not Completed | 7 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Moved to another state | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Withdrawal by clinical center | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs) | Total
Number analyzed (Participants) | 59 | 59 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment
  years | 10.2 (1.1) | 10.0 (1.1) | 10.1 (1.1)
Age, Customized [Number; unit: participants] — Age at enrollment
  participants
    8 to <9 years | 8 | 14 | 22
    9 to <10 years | 15 | 17 | 32
    10 to <11 years | 18 | 14 | 32
    11 to <12 years | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 23 | 31 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28 | 31 | 59
  African American | 14 | 10 | 24
  Hispanic or Latino | 10 | 12 | 22
  Asian | 5 | 4 | 9
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 59 | 59 | 118
Spectacle wear (single vision lenses) [Number; unit: participants]
  Currently | 33 | 33 | 66
  In past but not currently | 4 | 2 | 6
  Never | 22 | 24 | 46
Average Spherical Equivalent Between the Eyes [Number; unit: participants] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder and axis. In this study, sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle from 0 to 180 degrees (axis). Spherical equivalent is defined as the sphere plus 1/2 the cylinder. A spherical equivalent was calculated for each eye for each of the five trials of cycloplegic autorefraction, and the median for each eye was averaged to obtain the spherical equivalent used for analysis.
  participants
    -0.75 to -0.99 diopters (D) | 8 | 12 | 20
    -1.00 to -1.49 D | 22 | 23 | 45
    -1.50 to -1.99 D | 18 | 14 | 32
    -2.00 to -2.50 D | 11 | 10 | 21
Average Spherical Equivalent Between the Eyes [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. In this study, sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle from 0 to 180 degrees (axis). Spherical equivalent is defined as the sphere plus 1/2 the cylinder. A spherical equivalent was calculated for each eye for each of the five trials of cycloplegic autorefraction, and the median for each eye was averaged to obtain the spherical equivalent used for analysis.
  diopters | -1.50 (0.45) | -1.45 (0.47) | -1.48 (0.46)
Average J0 Between the Eyes [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. In this study, sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle from 0 to 180 degrees (axis). The dioptric power of a Jackson cross cylinder with axis at 0 degrees (J0) is calculated using the power vector approach. A J0 was calculated for each eye for each of the five trials of cycloplegic autorefraction, and the median for each eye was averaged to obtain the J0 used for analysis.
  diopters | -0.02 (0.18) | -0.02 (0.15) | -0.02 (0.16)
Average J45 Between the Eyes [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. In this study, sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle from 0 to 180 degrees (axis). The dioptric power of a Jackson cross cylinder with axis at 45 degrees (J45) is calculated using the power vector approach. A J45 was calculated for each eye for each of the five trials of cycloplegic autorefraction, and the median for each eye was averaged to obtain the J45 used for analysis.
  diopters | 0.11 (0.07) | 0.10 (0.07) | 0.11 (0.07)
Anisometropia [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. In this study, sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle from 0 to 180 degrees (axis). Anisometropia is defined as spherical equivalent in the right eye subtracted by spherical equivalent in the left eye.
  diopters | 0.22 (0.20) | 0.21 (0.16) | 0.22 (0.18)
Near Esophoria [Number; unit: participants] — Measured in prism diopters (PD) using the Prism and Alternate Cover Test (PACT) at 33 cm. Esophoria is the tendency of the eyes to deviate inwards when fusion between the eyes is suspended. Near esophoria is an esophoria when viewing close objects.
  participants
    2 to 5 prism diopters (PD) | 33 | 34 | 67
    6 to 10 PD | 22 | 21 | 43
    11 to 15 PD | 3 | 3 | 6
    16 to 20 PD | 1 | 1 | 2
Near Esophoria [Mean (Standard Deviation); unit: prism diopters] — Measured in prism diopters (PD) using the Prism and Alternate Cover Test (PACT) at 33 cm. Esophoria is the tendency of the eyes to deviate inwards when fusion between the eyes is suspended. Near esophoria is an esophoria when viewing close objects.
  prism diopters | 5.8 (3.2) | 5.9 (3.4) | 5.9 (3.3)
Accommodative Lag [Number; unit: participants] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle (axis). Accommodative lag is the average of the median accommodative lag of the five trials of the right eye. To determine the accommodative lag or accommodative lead, the accommodative measurement was added to the 3.00-D demand to result in the accommodative lag or lead. If the value was positive, it indicated accommodative lag; if the number was negative, it indicated accommodative lead.
  participants
    0.50 to 0.99 diopters (D) | 8 | 6 | 14
    1.00 to 1.49 D | 26 | 33 | 59
    1.50 to 1.99 D | 13 | 16 | 29
    2.00 D or more | 12 | 4 | 16
Accommodative Lag [Mean (Standard Deviation); unit: diopters] — Measured in diopters (D) using cycloplegic refraction sphere, cylinder, and axis. Sphere refers to the amount of myopia (nearsightedness) and cylinder the amount of astigmatism at a particular angle (axis). Accommodative lag is the average of the median accommodative lag of the five trials of the right eye. To determine the accommodative lag or accommodative lead, the accommodative measurement was added to the 3.00-D demand to result in the accommodative lag or lead. If the value was positive, it indicated accommodative lag; if the number was negative, it indicated accommodative lead.
  diopters | 1.47 (0.53) | 1.40 (0.48) | 1.44 (0.50)
Parental History of Myopia [Number; unit: participants]
  Neither parent | 10 | 5 | 15
  One parent | 16 | 10 | 26
  Both parents | 18 | 20 | 38
  Missing/unknown | 15 | 24 | 39

OUTCOME MEASURES:

1. Secondary Outcome: Distribution of Spherical Equivalent Refractive Error at 3 Years
Description: Measured in diopters (D) using cycloplegic refraction sphere (amount of myopia) and cylinder (amount of astigmatism at an angle (axis)). Spherical equivalent (SE) is defined as the sphere plus 1/2 the cylinder. A SE was calculated for each eye for each of the five trials of cycloplegic autorefraction, and the median for each eye was averaged to obtain the SE used for analysis.
Time Frame: 3 years
Population: The analysis followed the intent-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 52 | 58
participants
  Better than or equal to -0.49 D | 0 | 1
  -0.50 to -0.99 D | 2 | 1
  -1.00 to -1.99 D | 18 | 14
  -2.00 to -2.99 D | 20 | 21
  -3.00 to -3.99 D | 8 | 17
  Worse than or equal to -4.00 D | 4 | 4

2. Primary Outcome: Distribution of Change in Spherical Equivalent Refractive Error From Baseline to 3 Years
Description: Measured in diopters (D) using cycloplegic refraction sphere (amount of myopia) and cylinder (amount of astigmatism at an angle (axis)). Spherical equivalent (SE) is the sphere plus 1/2 the cylinder. For baseline and each time point, a SE was calculated for each eye for each of the five trials of cycloplegic autorefraction; the median for each eye was averaged to obtain the SE used for analysis. Change was calculated as SE at baseline minus SE at 3 years. A negative value indicates that the myopia worsened; a positive value indicates that it improved.
Time Frame: Baseline to 3 years
Population: The analysis followed the intent-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 52 | 58
participants
  >0.00 D (less myopia) | 6 | 3
  0.00 to -0.49 D | 11 | 8
  -0.50 to -0.99 D | 16 | 13
  -1.00 to -1.49 D | 12 | 13
  <= -1.50 D (more myopia) | 7 | 21

3. Secondary Outcome: Mean Spherical Equivalent Refractive Error at 3 Years
Description: as for outcome 1
Time Frame: 3 years
Population: The analysis followed the intent-to-treat principle.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 52 | 58
diopters | -2.41 (0.95) | -2.60 (0.91)

4. Primary Outcome: Mean Change in Spherical Equivalent Refractive Error From Baseline to 3 Years
Description: Measured in diopters (D) using cycloplegic refraction sphere (amount of myopia) and cylinder (amount of astigmatism at an angle (axis)). Spherical equivalent (SE) is defined as the sphere plus 1/2 the cylinder. For baseline and each time point, a SE was calculated for each eye for each of the five trials of cycloplegic autorefraction; the median for each eye was averaged to obtain the SE used for analysis. Change was calculated as SE at baseline minus SE at 3 years. A negative value indicates that the myopia worsened; a positive value indicates that it improved.
Time Frame: 3 years
Population: All analyses followed the intent-to-treat principle. The Monte Carlo Markov Chain (MCMC) method of multiple imputation was used to impute data for subjects who did not complete the 3-year visit.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 52 | 58
diopters | -0.87 (0.72) | -1.15 (0.75)
Statistical Analysis 1: Comparison: Progressive Addition Lenses (PALs) vs Single Vision Lenses (SVLs); The primary analysis was a comparison of treatment groups using an analysis of covariance (ANCOVA) model in which myopia at 3 years was adjusted for myopia at baseline and prior SVL wear. The sample size was computed to reach a 90% power and type I error rate of 5%, so that a difference in 3-year myopia progression between treatment groups would be detected if the true difference was at least 0.60 D, assuming a standard deviation of 0.85 D in each group and loss of follow up of 10%; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.28, 95% CI 2-sided [0.01 to 0.55]
Statistical Analysis 2: Comparison: Progressive Addition Lenses (PALs) vs Single Vision Lenses (SVLs); An adjusted analysis for the treatment group difference of change in spherical equivalent from baseline to 3 years was performed by including in an analysis of covariance (ANCOVA) model the following covariates in addition to baseline myopia and prior single vision lens wear, which are known to be related to myopia progression: age, sex, ethnicity, accommodative lag, and magnitude of near esophoria; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.27, 95% CI 2-sided [0.02 to 0.53]

5. Secondary Outcome: Distribution of Change in Spherical Equivalent Refractive Error From Baseline to 3 Years According to Baseline Characteristics
Description: Measured in diopters (D) using cycloplegic refraction sphere (amount of myopia) and cylinder (amount of astigmatism at an angle (axis)). Spherical equivalent (SE) is defined as the sphere plus 1/2 the cylinder. For baseline and 3 years, a SE was calculated for each eye for each of the five trials of cycloplegic autorefraction; the median for each eye was averaged to obtain the SE used for analysis. Change was calculated as SE at baseline minus SE at 3 years. A negative value indicates that the myopia worsened; a positive value indicates that it improved.
Time Frame: Baseline to 3 years
Population: The analysis followed the intent-to-treat principle.
Measure: Number; unit: participants
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 52 | 58
participants
  Age at baseline: 8 to <9 years | 8 | 13
  Age at baseline: 9 to <10 years | 13 | 17
  Age at baseline: 10 to <11 years | 15 | 14
  Age at baseline: 11 to <12 years | 16 | 14
  Gender: Male | 19 | 31
  Gender: Female | 33 | 27
  Race/Ethnicity: White | 26 | 30
  Race/Ethnicity: Nonwhite | 26 | 28
  Prior spectacle wear: Currently or in past | 31 | 34
  Prior spectacle wear: Never | 21 | 24
  Spherical equivalent at baseline: -0.75 to -1.49 D | 25 | 33
  Spherical equivalent at baseline: -1.50 to -2.50 D | 27 | 25
  Accommodative lag at baseline: 0.50 to 1.49 D | 28 | 38
  Accommodative lag at baseline: 1.50 or worse | 24 | 20
  Near esophoria at baseline: 2 to 5 PD | 30 | 33
  Near esophoria at baseline: 6 to 10 PD | 18 | 21
  Near esophoria at baseline: >10 PD | 4 | 4
  Parental history of myopia: Neither parent | 9 | 5
  Parental history of myopia: One parent | 15 | 10
  Parental history of myopia: Both parents | 18 | 20

6. Secondary Outcome: Mean Change in Spherical Equivalent Refractive Error From Baseline to 3 Years According to Baseline Characteristics
Description: as for outcome 5
Time Frame: Baseline to 3 years
Population: The analysis followed the intent-to-treat principle.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 52 | 58
diopters
  Age at baseline: 8 to <9 years | -1.23 (1.06) | -1.39 (0.79)
  Age at baseline: 9 to <10 years | -1.11 (0.76) | -1.14 (0.78)
  Age at baseline: 10 to <11 years | -0.71 (0.52) | -1.19 (0.81)
  Age at baseline: 11 to <12 years | -0.64 (0.55) | -0.88 (0.58)
  Gender: Male | -0.95 (0.64) | -1.09 (0.75)
  Gender: Female | -0.82 (0.76) | -1.21 (0.76)
  Race/Ethnicity: White | -0.79 (0.74) | -1.10 (0.76)
  Race/Ethnicity: Nonwhite | -0.94 (0.70) | -1.19 (0.75)
  Prior spectacle wear: Currently or in past | -0.90 (0.75) | -1.10 (0.63)
  Prior spectacle wear: Never | -0.81 (0.68) | -1.22 (0.90)
  Spherical equivalent at baseline: -0.75 to -1.49 D | -0.79 (0.61) | -1.20 (0.76)
  Spherical equivalent at baseline: -1.50 to -2.50 D | -0.93 (0.81) | -1.08 (0.75)
  Accommodative lag at baseline: 0.50 to 1.49 D | -0.91 (0.59) | -1.12 (0.72)
  Accommodative lag at baseline: 1.50 or worse | -0.81 (0.86) | -1.20 (0.82)
  Near esophoria at baseline: 2 to 5 PD | -0.97 (0.82) | -1.13 (0.79)
  Near esophoria at baseline: 6 to 10 PD | -0.66 (0.54) | -1.09 (0.67)
  Near esophoria at baseline: >10 PD | -1.01 (0.43) | -1.60 (0.86)
  Parental history of myopia: Neither parent | -0.83 (0.63) | -0.72 (0.76)
  Parental history of myopia: One parent | -0.73 (0.52) | -1.28 (0.62)
  Parental history of myopia: Both parents | -0.99 (0.79) | -1.29 (0.87)

7. Secondary Outcome: Mean Change in Spherical Equivalent Refractive Error From Baseline to 1 Year
Description: Measured in diopters (D) using cycloplegic refraction sphere (amount of myopia) and cylinder (amount of astigmatism at an angle (axis)). Spherical equivalent (SE) is defined as the sphere plus 1/2 the cylinder. For baseline and 1 year, a SE was calculated for each eye for each of the five trials of cycloplegic autorefraction; the median for each eye was averaged to obtain the SE used for analysis. Change was calculated as SE at baseline minus SE at 1 year. A negative value indicates that the myopia worsened; a positive value indicates that it improved.
Time Frame: Baseline to 1 year
Population: The analysis followed the intent-to-treat principle.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 55 | 58
diopters | -0.29 (0.39) | -0.42 (0.37)
Statistical Analysis 1: Comparison: Progressive Addition Lenses (PALs) vs Single Vision Lenses (SVLs); A secondary analysis was conducted to assess the treatment effect on myopia at the interim time point of 1 year, using an analysis of covariance (ANCOVA) model for the treatment group difference of change in spherical equivalent refractive error from baseline to 1 year, in which myopia at 1 year was adjusted for myopia at baseline and prior single vision lenses wear. Only complete cases (cases in which both baseline and 1 year values were known) were included; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.005 to 0.28]

8. Secondary Outcome: Mean Change in Spherical Equivalent Refractive Error From Baseline to 2 Years
Description: Measured in diopters (D) using cycloplegic refraction sphere (amount of myopia) and cylinder (amount of astigmatism at an angle (axis)). Spherical equivalent (SE) is defined as the sphere plus 1/2 the cylinder. For baseline and 2 years, a SE was calculated for each eye for each of the five trials of cycloplegic autorefraction; the median for each eye was averaged to obtain the SE used for analysis. Change was calculated as SE at baseline minus SE at 2 years. A negative value indicates that the myopia worsened; a positive value indicates that it improved.
Time Frame: Baseline to 2 years
Population: The analysis followed the intent-to-treat principle
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 55 | 58
diopters | -0.58 (0.55) | -0.80 (0.61)
Statistical Analysis 1: Comparison: Progressive Addition Lenses (PALs) vs Single Vision Lenses (SVLs); A secondary analysis was conducted to assess the treatment effect on myopia at the interim time point of 2 years, using an analysis of covariance (ANCOVA) model for the treatment group difference of change in spherical equivalent refractive error from baseline to 2 years, in which myopia at 2 years was adjusted for myopia at baseline and prior single vision lenses wear. Only complete cases (cases in which both baseline and 2 year values were known) were included; Test type: Superiority or Other; ANCOVA; Mean Difference (Net) = 0.23, 95% CI 2-sided [0.02 to 0.45]

9. Secondary Outcome: Excellent Spectacle Compliance
Description: Spectacle compliance was assessed on a five-point Likert scale: always, 5; often, 4; sometimes, 3; rarely, 2; and never, 1. Excellent compliance indicates that for the specified period (during school, after school, on weekends), spectacles were estimated at all visits to have been worn either always or often.
Time Frame: Baseline to 3 years
Population: The analysis followed the intent-to-treat principle. Two patients had no compliance data because they had no follow-up visits (one single vision lenses, and one progressive-addition lenses).
Measure: Number; unit: percent of participants
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Number analyzed (Participants) | 58 | 58
percent of participants
  During school | 72 | 90
  After school | 60 | 76
  Weekends | 60 | 71

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 3-year outcome visit.
Arm/Group | Progressive Addition Lenses (PALs) | Single Vision Lenses (SVLs)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59

LIMITATIONS AND CAVEATS:
Limitations include: differential loss to follow up , differential compliance between the groups, power of near addition was not customized in PAL group, and we have no data on whether PAL group was looking through the near addition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No